CLINICAL TRIAL: NCT05496569
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase II Clinical Trial of TQB3616 Capsules Versus Placebo in the Treatment of Dedifferentiated Liposarcoma
Brief Title: TQB3616 Capsules in the Treatment of Dedifferentiated Liposarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was closed due to business reasons. Closure was not prompted by any safety or efficacy concerns.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TQB3616-II-03（stage2）
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-09

CONDITIONS: Dedifferentiated Liposarcoma
MeSH Terms: conditions — Liposarcoma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB3616 capsules (Experimental): TQB3616 capsule (180mg, quaque die, oral), 4 weeks (28 days) as a treatment cycle.
  Interventions: Drug: TQB3616 capsule
- TQB3616 placebo (Placebo Comparator): TQB3616 placebo (0mg, quaque die, oral), 4 weeks (28 days) as a treatment cycle.
  Interventions: Drug: TQB3616 placebo

INTERVENTIONS:
Drug: TQB3616 capsule — TQB3616 capsule is a cyclin-dependent kinase 4/6 kinase inhibitor
  Arms: TQB3616 capsules
Drug: TQB3616 placebo — Placebo
  Arms: TQB3616 placebo

SUMMARY:
A clinical trial evaluating TQB3616 capsules versus placebo in the treatment of dedifferentiated liposarcoma. Divided into 2 stages, the second stage, a total of 118 subjects are planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 1 Subjects shall voluntarily join the research, capable of giving written informed consent with good compliance;
* 2 Age: 18-75 years old (calculated based on the time of signing the informed consent form); The Eastern Cooperative Oncology Group performance status (ECOG PS) score: 0-1 points; Body mass index (BMI)>18.5 and body weight>40kg; Expected survival time>3 months;
* 3 Patients with dedifferentiated liposarcoma who were diagnosed as unresectable or refused surgery after multidisciplinary consultation, and the pathological and imaging review results showed the presence of dedifferentiated liposarcoma component, and the subjects must also meet any of the following categories:

  1. Newly diagnosed dedifferentiated liposarcoma;
  2. Patients with residual disease after surgery;
  3. Local recurrence and metastatic dedifferentiated liposarcoma;
  4. Patients with disease progression confirmed by imaging results within nearly 6 months; Note: Difficult to resection by surgery: （R0：Complete tumor resection /R1：Residual tumor cells at the resection margin ）resection cannot be achieved by surgery according to the investigator's assessment: ①The tumor is huge or involves important organs; ②The tumor is located in an important vascular pathway; ③The tumor has multiple metastases, It is difficult to control by surgery; ④ Combination of serious medical diseases can cause fatal surgical risks; ⑤ Recurrence after multiple operations is not suitable for immediate surgery.

Treatment-naive subjects: Subjects who have not received systemic drug therapy or have not relapsed within 6 months after postoperative adjuvant therapy.

Treatment-experienced subjects: Subjects who have relapsed within 6 months after receiving first-line systemic drug therapy or postoperative adjuvant therapy.

* 4 According to the Response Evaluation Criteria in Solid Tumors 1.1（RECIST 1.1） criteria, there is at least one measurable lesion. If the measurable lesion is located in the area of previous radiotherapy, it should be clearly defined as a progressive state;
* 5 Subjects have recovered to ≤Grade 1 or baseline (according to Common Terminology Criteria for Adverse Events Version 5.0 [CTCAE v 5.0]), alopecia and peripheral Grade 2 all acute toxic effects of prior treatment or surgery prior to first dose except for neuropathy;
* 6 Adequate major organ function meeting the following criteria:

  1. Routine blood tests criteria (no blood transfusion or correction with hematopoietic stimulating factor drugs within 7 days before the examination):

     1. Hemoglobin (HGB)≥90.0g/L;
     2. Absolute neutrophil value (ANC)≥1.5×109/L;
     3. Platelet count (PLT)≥90×109/L;
  2. Biochemical examination criteria:

     1. Total bilirubin (TBIL)≤1.5 times the upper limit of normal (ULN); Gilbert syndrome patients≤3×ULN;
     2. Amino acid aminotransferase (ALT) and aspartate aminotransferase (AST)≤3×ULN. If accompanied by liver metastasis, ALT and AST≤5×ULN;
     3. Serum creatinine (CR)≤178μmol/L or creatinine clearance rate (CCR)>50ml/min;
  3. Urine routine examination criteria: Urine routine indicates urine protein<++; if urine protein≥++, the 24-hour urine protein quantification should be confirmed≤1.0 g;
  4. Coagulation function criteria: Prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio (INR)≤1.5×ULN (no anticoagulation therapy);
  5. Echocardiography assessment: Left ventricular ejection fraction (LVEF)≥50%;
  6. 12-lead Electrocardiogram（ECG）assessment: QTc<450ms (male), QTc<470ms (female).
* 7 Female subjects of childbearing age shall agree to use contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; serum pregnancy test negative within 7 days before study enrollment , and must be non-lactating subjects; male subjects shall agree to use contraception during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

* 1 Tumor disease and medical history:

  1. Subjects with atypical lipomatous tumor/well-differentiated liposarcoma, myxoid/round cell liposarcoma, pleomorphic liposarcoma on pathology and imaging review;
  2. Have developed or currently suffers from other malignant tumors within past 3 years. The following two conditions were eligible for enrollment: Other malignancies treated with single surgery, achieving 5 consecutive years of disease-free survival (DFS); Cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor-infiltrating basement membrane)]; Patients with other sources of carcinoma in situ and patients with previous malignancies who are currently in remission will be eligible to participate in the study if the investigator determines that the likelihood of recurrence is very low and will require sponsor approval prior to enrollment of these patients;
  3. Severe bone damage caused by tumor bone metastasis; including pathological fractures of weight-bearing bones (such as vertebrae, pelvis, femur, tibia, phalanges, calcaneus, etc.) and spinal cord compression that occurred within 6 months or that the investigators judged to be likely to occur in the near future;
  4. Imaging Computed Tomography or Magnetic Resonance Imaging (CT or MRI) shows the presence of tumor thrombus, brain metastasis or the number of lesions > 10;
  5. Uncontrolled pleural effusion, pericardial effusion or ascites that still needs repeated drainage (judgment by the investigator).
* 2 Previous anti-tumor or concomitant drug therapy:

  1. Received chemotherapy (including anthracyclines), radiotherapy, major surgery, biological therapy, cytokine immunotherapy, hormone therapy, clinical trial drug therapy, traditional Chinese medicine with anti-tumor indications or Chinese patent medicine, etc.
  2. Received major surgery, major surgical treatment, incisional biopsy, obvious traumatic injury within 4 weeks before the first treatment with the study drug, or has not been able to fully recover from the previous surgery as judged by the investigator, and has anti-tumor indications Chinese medicine or proprietary Chinese medicine, etc.;
  3. Previously received Abemaciclib or Palbociclib and any other CDK4/6 inhibitor treatment;
  4. The target drug (or anti- programmeddeath-1/ Programmed cell death 1 ligand 1 and other immune drugs) is not used for at least 5 half-lives (calculated from the end of the last treatment) from the time of first receiving the study drug to the last time. If it is a combination drug, calculated based on the drug with the longest half-life;
  5. After receiving the study drug for the first time subjects who have used drugs or traditional chinese medicines containing strong Cytochrome P450 3A4(CYP3A4) inhibitors or inducers (such as Carbamazepine, Phenobarbital, Pioglitazone, etc.) within the first 4 weeks and cannot be stopped during the treatment period;
* 3 Comorbid diseases and medical history:

  1. Liver abnormalities:

     1. Decompensated cirrhosis (Child-Pugh liver function Grade B or C);
     2. Active or chronic hepatitis (Hepatitis B reference: Hepatitis B Surface Antigen (HBsAg) positive, Hepatitis B Virus DeoxyriboNucleic Acid (HBV-DNA)>1000 copies/mL or>200IU/mL; Hepatitis C reference: Hepatitis C virus (HCV )antibody positive, and the HCV virus titer detection value exceeds the upper limit of the normal value); HBV surface antigen positive or core antibody positive, HCV antibody positive subjects who meet the entry conditions, after antiviral treatment subjects who meet the above criteria can be admitted into the group, and antiviral drugs can be used to prevent virus activation during the group period.
     3. Patients with ascites or bleeding diseases secondary to hepatic insufficiency.
  2. Renal abnormalities: renal failure requiring hemodialysis or peritoneal dialysis;
  3. Cardiovascular and cerebrovascular abnormalities:

     1. Patients with a history of epilepsy, or a history of seizures, disturbance of consciousness or transient ischemic attack within the last 12 months, or a history of unexplained coma;
     2. New York Heart Association Grade II to IV heart failure as defined by grade. Second degree or higher heart block, myocardial infarction or arterial thrombosis event, unstable arrhythmia or unstable angina pectoris within the past 6 months;
     3. Cerebrovascular accident, cerebral infarction, etc. occurred within 6 months;
     4. Hypertension uncontrolled by drugs (systolic blood pressure≥150mmHg, diastolic blood pressure≥100mmHg); For patients with a history of hypertension, if blood pressure is well controlled by antihypertensive therapy, they are allowed to participate in this study;
     5. Past or current heart valve inflammation, endocarditis;
     6. Cardiovascular syncope, pathological ventricular arrhythmia (including but not limited to ventricular tachycardia and ventricular fibrillation) or sudden cardiac death. Atrial fibrillation or other cardiac arrhythmia requiring medication.
  4. Gastrointestinal tract abnormalities:

     1. Inability to take oral medication (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.);
     2. History of malabsorption syndrome or other diseases that interfere with gastrointestinal absorption;
     3. Cerebrovascular accident, cerebral infarction, etc. occurred within 6 months;
     4. Chronic diarrhea of Grade 2 or above persists despite the maximum medical treatment;
     5. The investigator judged that it may cause gastrointestinal bleeding and perforation other conditions.
  5. Immunodeficiency history:

     1. Known human immunodeficiency virus (HIV) infection;
     2. Other acquired and congenital immunodeficiency diseases;
     3. Prepared or previously received organ transplantation, or received within 60 days before the first dose Hematopoietic stem cell transplantation, or with obvious host transplantation response (except corneal transplantation);
     4. Systemic or topical immunosuppressive or hormonal therapy is required to achieve immunosuppression, and glucocorticoids must continue to be used within 7 days before the first dose Hormones, or patients who still need to use immunosuppressive drugs within 5 half-lives before the first dose (daily dose of glucocorticoid <7.5 mg prednisone or other equivalent therapeutic hormones, autoimmune-related diseases judged by the investigator to be in stable phase) except patients).

     Note: Hormone replacement therapy (e.g., Tthyroxine, Insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered systemic therapy and is permitted.
  6. Bleeding risk:

     1. Suffering from bleeding (hemoptysis), coagulation disease, or using Warfarin, Aspirin and other antiplatelet agglutination drugs (except Aspirin ≤100 mg/d for prophylaxis);
     2. Regardless of severity, with any signs or history of bleeding constitution;
     3. Any CTCAE ≥ Grade 3 bleeding or bleeding events within 4 weeks prior to the first dose.
  7. The patients have an active systemic infection (such as a bacterial infection requiring intravenous antibiotic therapy at the start of study treatment, a fungal infection, or a detectable viral infection requiring systemic therapy) or an excessive viral load.
  8. History of idiopathic pulmonary fibrosis, history of organized pneumonia (e.g., bronchiolitis obliterans), history of drug-induced pneumonia, history of idiopathic pneumonia, or evidence of active pneumonia on chest CT scan during screening.
  9. There is a clear history of neurological or psychiatric disorders in the past.
  10. Combined with severe or uncontrolled diseases, the investigators judge that there may be a greater risk of entering this study, including but not limited to:

      1. Type 1 or type 2 diabetes that cannot be controlled by drugs (or fasting blood glucose (FBG) > 10mmol/L);
      2. Thyroid disease;
      3. Treponema pallidum specific antibody positive.
  11. Pituitary or adrenal dysfunction history.
  12. Received major surgical treatment, incisional biopsy or significant traumatic injury within 4 weeks prior to the start of study treatment.
  13. Long-term unhealed wounds or fractures.
  14. Subjects who have a drug abuse history and cannot quit or have a drug use history.
* 4 Study treatment related:

  1. Have a severe allergic disease, drug allergy history, or known allergy to the components of TQB3616 capsule and its adjuvants and similar drugs;
  2. Active autoimmune disease requiring systemic therapy (such as the use of disease-modifying drugs, corticosteroids, or immunosuppressive drugs) within 2 years prior to the start of study treatment (including but not limited to: autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis; asthma requiring bronchodilator medical intervention is not included);
* 5 Subjects judged by the investigator to have the possibility of recent rapid progress, need to receive chemotherapy or lack of compliance;
* 6 According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or there are subjects who are not suitable for enrollment for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2025-09-28 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by an independent review committee | 18 to 24 months
  From randomization to the time of disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Progression-free survival assessed by the investigator. | 14 to 24 months
  From randomization to the time of disease progression or death, whichever occurs first.
Overall survival | 20 to 30 months
  From randomization to the time of death from any cause.
Duration of disease remission | 18 to 24 months
  For subjects whose best remission is complete remission or partial remission , it is defined as from the date when tumor remission is first recorded to the date when disease progression is first recorded or the date of death from any cause, whichever occurs first.
Objective response rate | 24 months
  Percentage of complete or partial remission subjects as determined by RECIST 1.1.
Disease control rate | 24 months
  Percentage of subjects with complete remission, partial remission, or disease stabilization at 6 weeks or more as determined by RECIST 1.1.
Progression-free survival after crossover in control subjects | 18 to 30months
  From the beginning of the crossover to the time of disease progression or death, whichever is first discovered
Adverse events , abnormal laboratory values, and serious adverse events | 27 months
  All adverse medical events that occurred after the subject received the investigational drug.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality